CLINICAL TRIAL: NCT04058522
Title: Treatment of Subacromial Shoulder Pain by Individual or Group Physiotherapy Following Corticosteroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Eastern Health and Social Care Trust (Other)
Collaborators: Northern Ireland Clinical Trials Unit (Other); University of Ulster (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Ian Ryans, General Practitioner, South Eastern Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10.05.7
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Shoulder Pain; Rotator Cuff Impingement
Keywords: Physiotherapy; Group Treatment
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Single blind randomised trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Off site randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Physiotherapy (Experimental): 1 class per week for 6 weeks (30 min length) aiming for 5-10 participants per class. Classes included advice on the nature of the condition and exercises for scapulo-humeral mobility, scapulo-humeral stability and specific rotator cuff rehabilitation exercises
  Interventions: Other: Rotator cuff rehabilitation classes; Drug: Triamcinolone Injection
- Routine Physiotherapy (Active Comparator): Individual physiotherapy sessions: 6 sessions weekly (30 min) for 6 weeks. Treatment was based on evidence-based guidelines for the treatment of shoulder impingement (CSP 2005) and consisted of mobilisation techniques, supervised exercises and stretches.
  Interventions: Other: Individual Physiotherapy; Drug: Triamcinolone Injection

INTERVENTIONS:
Other: Rotator cuff rehabilitation classes
  Arms: Group Physiotherapy
Other: Individual Physiotherapy
  Arms: Routine Physiotherapy
Drug: Triamcinolone Injection — Subacromial Injection 40mg/1ml
  Other Names: Kenalog Injection

SUMMARY:
The aim of this study is therefore to examine the clinical effectiveness and provide an economic analysis of individual versus group physiotherapy, following corticosteroid injection, for management of Subacromial Impingement (SAI) of the shoulder.

DETAILED DESCRIPTION:
This trial was a single blind, randomised, equivalence trial comparing rotator cuff rehabilitation classes with traditional individual physiotherapy in subacromial impingement of the shoulder. A total of 200 patients were planned to be recruited from patients with painful shoulder referred to the Ulster Community and Hospitals Trust and community physiotherapy at the Ulster, Ards and Bangor sites or injection clinics at the Ulster Hospital. Local General Practitioners were also informed of the study and invited to refer appropriate patients.

Intervention - Triamcinolone 40 mg (1 ml) and 6 weekly rotator cuff rehabilitation classes Control - Triamcinolone 40 mg (1 ml) and routine physiotherapy 6 sessions weekly for 6 weeks

The injection technique involving a lateral approach to the subacromial space was used. An interval of between 1 and 3 weeks was allowed between injection and commencement of classes or physiotherapy.

Classes were planned to be run by a rotating group of physiotherapists with at least 1 year of musculoskeletal outpatient's experience. They were to receive instruction on the protocol to use in the classes. Classes were to consist of six 30 min sessions on a weekly basis. A minimum of 5 and maximum of 10 participants were to attend. Advice was to be given on the nature of the condition. Subjects were to be instructed and supervised in exercises for scapulo-humeral mobility, scapulo-humeral stability and specific rotator cuff rehabilitation exercises. Subjects were to be introduced to ongoing classes as they are recruited to the trial.

Six sessions of routine physiotherapy at weekly intervals were to be undertaken. Treatment was to be based on evidence-based guidelines for the treatment of shoulder impingement (Evidence-based clinical guidelines for the diagnosis, assessment and physiotherapy management of shoulder impingement syndrome Chartered Society of Physiotherapists 2005) and consist of mobilisation techniques and supervised exercises and stretches. A therapist with at least 1 year of musculoskeletal outpatients experience was to provide treatments.

ELIGIBILITY:
Inclusion Criteria:

* unilateral shoulder pain of more than 4 weeks duration and a Shoulder Pain and Disability Index (SPADI) score of >= 30 as this represents significant disability. Shoulder pain is defined as pain in the shoulder region, including the upper arm, elicited by active or passive shoulder movement. The diagnosis of "subacromial pain" is defined by range as no limitation in passive range of movement or restriction of passive range of movement mainly in abduction rather than external rotation.

Exclusion Criteria:

* inability to give informed consent
* physiotherapy or injection treatment for current shoulder pain in previous 3 months
* blood coagulation disorders
* bilateral shoulder pain
* evidence of systemic infection
* abnormal shoulder X-ray defined as significant glenohumeral or subacromial joint space narrowing suggesting osteoarthritis of glenohumeral joint or complete rotator cuff rupture,
* evidence of rotator cuff tear, tested by external rotation lag sign, drop sign, internal rotation lag sign and static muscle resistance in external rotation, internal rotation and abduction,
* history of significant trauma to the shoulder,
* inflammatory joint disease,
* history of cerebrovascular accident,
* allergy or contraindication to Triamcinolone/contraindication to injection.
* evidence of referred pain from cervical spine disease.
* pregnancy or breast feeding
* patients whose first language is not English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2013-02-10 (Actual); Study Completion 2013-02-10 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index (SPADI) | 26 Weeks
  The shoulder pain and disability index

SECONDARY OUTCOMES:
Active range of external rotation | 26 weeks
  Range of active external rotation of the shoulder measured by goniometer.
Internal rotation | 26 weeks
  Measures as distance in centimetres between thumb tip and C7 spinous process)
Global patient self-assessment | 26 weeks
  Self assessment of global wellbeing measured by a 100mm visual analogue scale. Score minimum 0 and maximum 100 higher score indicates higher wellbeing.
Short Form 36 version 2 (SF36v2) | 26 weeks
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are, vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.
  Each scale is transformed into a 0-100 scale. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
EuroQuol 5 - Dimensions - 3 Levels (EQ-5D-3L) | 26 weeks
  EuroQol's EQ-5D is a generic instrument to measure and evaluate health status. The EQ-5D 3L version, describes general health based on five distinct dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 Levels (indicating no problem, some or moderate problem and extreme problem). EQ-5D comprises of five domains, each with three possible levels, a combination of the characteristic levels produces 243 possible health states (ranging from 11111 to 33333). The EQ-5D index scores are utilities derived from the respondents profile and ranges from 0 to 1; 0 meaning death and 1 complete health.
Hospital Anxiety and Depression Scale (HADS) | 26 weeks
  The HAD questionnaire comprises seven questions for anxiety and seven questions for depression. The anxiety and depression questions are interspersed within the questionnaire but are scored separately. Cut-off scores are available for quantification, for example a score of 8 or more for anxiety has a specificity of 0.78 and a sensitivity of 0.9, and for depression a specificity of 0.79 and a sensitivity of 0.83. Each scale has a range of 0-21. Scores of 15-21 indicate severe, 11-14, moderate and 8-10 mild, 7 or less indicates no case

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ryans, MD, Principal Investigator — Dundonald Medical Centre
Locations (1):
- Ian Ryans, Dundonald, Co Down, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryans I, Galway R, Harte A, Verghis R, Agus A, Heron N, McKane R. The Effectiveness of Individual or Group Physiotherapy in the Management of Sub-Acromial Impingement: A Randomised Controlled Trial and Health Economic Analysis. Int J Environ Res Public Health. 2020 Aug 1;17(15):5565. doi: 10.3390/ijerph17155565. PMID 32752234